CLINICAL TRIAL: NCT02770482
Title: Utility of Amyloid Beta-peptide 1-40 Measurement in the Diagnosis of Alzheimer's Disease
Brief Title: Amyloid Beta-peptide 1-40 and Alzheimer's Disease
Acronym: ADAB40
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA13050
Record Dates: First submitted 2015-03-31; First posted 2016-05-12 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer Disease
Keywords: dementia; biomarkers; cerebrospinal fluid
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AD Patients (Experimental)
  Interventions: Biological: spinal fluid collection

INTERVENTIONS:
Biological: spinal fluid collection

SUMMARY:
The combined measurement of Ab42 and tau protein (total and phosphorylated) in the spinal fluid has been shown to be promising in the diagnosis of Alzheimer's disease (AD), and has justified its inclusion new diagnostic criteria. However, it can sometimes yield discordant results that are not discriminant (isolated variation in Ab42 or P-181 Tau). To answer this challenge, a new marker has been developed in recent years, namely amyloid beta-peptide 1-40 (Aβ40). This marker reflects the patient's total amyloid deposits and is used to calculate the Aβ42/Aβ40 ratio. This ratio measures the relative variation of Aβ42 as compared to the total amyloid burden. Literature data on this topic are sparse and to date, no report has been published evaluating the utility of this marker in the diagnostic strategy for AD.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the Memory Clinic of Champagne-Ardennes for memory disorders, and
* Whose diagnostic work-up requires assessment of biomarkers present in the cerebrospinal fluid are considered eligible for inclusion in this study.

Exclusion Criteria:

* Patients who do not have any social security coverage will not be included.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-06; Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Percentage of diagnostic certitude for AD (diagnosed cases) | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Background] Kisserli A, Tabary T, Cohen JHM, Duret V, Mahmoudi R. High-resolution Melting PCR for Complement Receptor 1 Length Polymorphism Genotyping: An Innovative Tool for Alzheimer's Disease Gene Susceptibility Assessment. J Vis Exp. 2017 Jul 18;(125):56012. doi: 10.3791/56012. PMID 28745649